CLINICAL TRIAL: NCT02250430
Title: A Phase 1, Single-Center, Split-Face Study Assessing Local Cutaneous Effects After Application of SB204 2% and SB204 4% in Healthy Volunteers
Brief Title: A Phase 1 Study Assessing Local Cutaneous Effects of SB204
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-AC102
Record Dates: First submitted 2014-09-10; First posted 2014-09-26 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Acne Vulgaris
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topical SB204 (Experimental): Topical application of SB204 2% and 4% twice daily for 2 days and once on Day 3
  Interventions: Drug: SB204

INTERVENTIONS:
Drug: SB204 — Applied topically twice a day on days 1, 2 and 3 to left and right cheeks
  Other Names: NVN1000

SUMMARY:
In this study, color (erythema) and pH will be measured on 3 consecutive days after application of 2 doses of SB204 to the cheeks of healthy volunteers.

DETAILED DESCRIPTION:
This study is to evaluate local cutaneous effects, including intensity and duration of erythema and changes in pH following 5 applications (twice daily for two days and once daily on the third day) of SB204 2% and SB204 4% twice daily to the face for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Women who are pregnant or nursing
* Subject with known sensitivity to a component of the test materials

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Intensity of erythema following application of SB204 2% and SB204 4%. | 3 days
Duration of erythema following application of SB204 2% and SB204 4%. | 3 days

SECONDARY OUTCOMES:
pH on the surface of the skin after topical application of 2 concentrations of SB204 | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Lessin, MD, Principal Investigator — KGL, Inc.
Locations (1):
- KGL, Broomall, Pennsylvania, United States